CLINICAL TRIAL: NCT01807000
Title: A Phase 1 Study to Investigate the Absorption, Metabolism, and Excretion of [14C] Prucalopride Succinate Following a Single Oral Dose in Healthy Male Subjects
Brief Title: Absorption, Metabolism and Excretion (AME) of Single Dose Radiolabeled Prucalopride Succinate in Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SPD555-104
Record Dates: First submitted 2013-03-06; First posted 2013-03-08 (Estimated); Results first posted 2014-09-05 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiolabeled Prucalopride Succinate (Experimental)
  Interventions: Drug: Radiolabeled Prucalopride Succinate

INTERVENTIONS:
Drug: Radiolabeled Prucalopride Succinate — A single oral dose of 2 mg radiolabeled prucalopride succinate administered on Day 1.

SUMMARY:
Phase I study to evaluate the excretion of radioactivity, the metabolic profile, pharmacokinetics, safety and tolerability following a single oral administration of [14C] Prucalopride Succinate in healthy male volunteers aged 18 to 50 years (inclusive).The purpose of this study is to investigate how and how quickly Prucalopride Succinate or its break down products are excreted by analysing blood, faeces and urine samples collected during the study.

ELIGIBILITY:
Inclusion Criteria:

* Males aged between 18 and 50 years, inclusive
* Body mass index (BMI) of ≥18 and ≤30 kg/m2
* No more than 2 bowel movements per day or fewer than 3 bowel movement per week
* Provision of signed and dated, written informed consent prior to any study specific procedures

Exclusion Criteria:

* Have participated in a [14C]-study within the last 6 months.
* Exposure to clinically significant radiation within 12 months prior to dose (for example, serial X-ray or computed tomography scans, barium meal, current employment in a job requiring radiation exposure monitoring).
* Male subjects who consume more than 21 units of alcohol per week or 3 units per day.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2013-03-18 (Actual); Primary Completion 2013-04-28 (Actual); Study Completion 2013-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Covance Global Clinical Research Unit Inc., Madison, Wisconsin, United States

REFERENCES:
- [Derived] Flach S, Scarfe G, Dragone J, Ding J, Seymour M, Pennick M, Pankratz T, Troy S, Getsy J. A Phase I Study to Investigate the Absorption, Pharmacokinetics, and Excretion of [(14)C]Prucalopride After a Single Oral Dose in Healthy Volunteers. Clin Ther. 2016 Sep;38(9):2106-15. doi: 10.1016/j.clinthera.2016.08.003. Epub 2016 Sep 7. PMID 27614912

RESULTS

PARTICIPANT FLOW:
Groups:
- [14C] PRUCALOPRIDE SUCCINATE: A single oral dose of 2 mg radiolabeled prucalopride succinate administered on Day 1.
Period: Overall Study
Arm/Group | [14C] PRUCALOPRIDE SUCCINATE
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | [14C] PRUCALOPRIDE SUCCINATE
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.5 (10.45)
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 6

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to Infinity (AUC 0→∞) of Radiolabelled Prucalopride Succinate
Description: AUC can be used as a measure of drug exposure. It is derived from drug concentration and time so it gives a measure how much and how long a drug stays in a body.
Time Frame: Over 240 hours post-dose
Population: The Pharmacokinetic Analysis Set included all subjects with at least 1 pharmacokinetic parameter estimated adequately in the Pharmacokinetic Concentration Analysis Set which included all subjects who took 1 dose of investigational product, underwent plasma pharmacokinetic sampling, and had evaluable pharmacokinetic assay results.
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | [14C] PRUCALOPRIDE SUCCINATE
Number analyzed (Participants) | 6
ng*h/ml | 96.5 (9.64)

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of Radiolabelled Prucalopride Succinate
Description: Cmax is a term that refers to the maximum (or peak) concentration that a drug achieves in the body after the drug has been administered.
Time Frame: Over 240 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | [14C] PRUCALOPRIDE SUCCINATE
Number analyzed (Participants) | 6
ng/ml | 3.79 (1.10)

3. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) of Radiolabelled Prucalopride Succinate
Description: Tmax is the time after administration of a drug when the maximum plasma concentration in the body is reached.
Time Frame: Over 240 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Median (Full Range); unit: hours
Arm/Group | [14C] PRUCALOPRIDE SUCCINATE
Number analyzed (Participants) | 6
hours | 2.75 [1.13 to 4.00]

4. Primary Outcome: Plasma Half-Life (T1/2) of Radiolabelled Prucalopride Succinate
Description: The time it takes for the blood plasma concentration of a substance to halve.
Time Frame: Over 240 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | [14C] PRUCALOPRIDE SUCCINATE
Number analyzed (Participants) | 6
hours | 20.6 (5.35)

5. Primary Outcome: Total Body Clearance (CL/F) of Radiolabelled Prucalopride Succinate
Description: The rate at which a drug is removed from the body.
Time Frame: Over 240 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | [14C] PRUCALOPRIDE SUCCINATE
Number analyzed (Participants) | 6
L/h | 20.9 (2.07)

6. Primary Outcome: Volume of Distribution (Vz/F) of Radiolabelled Prucalopride Succinate
Description: The distribution of a medication between plasma and the rest of the body.
Time Frame: Over 240 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | [14C] PRUCALOPRIDE SUCCINATE
Number analyzed (Participants) | 6
Liters | 623 (185)

7. Primary Outcome: AUC 0→∞ Whole Blood Total Radioactivity of Radiolabelled Prucalopride Succinate
Time Frame: Over 240 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: ng equivalents*h/ml
Arm/Group | [14C] PRUCALOPRIDE SUCCINATE
Number analyzed (Participants) | 6
ng equivalents*h/ml | 192 (31.9)

8. Primary Outcome: Cmax Whole Blood Total Radioactivity of Radiolabelled Prucalopride Succinate
Time Frame: Over 240 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: ng equivalents/ml
Arm/Group | [14C] PRUCALOPRIDE SUCCINATE
Number analyzed (Participants) | 6
ng equivalents/ml | 7.74 (2.34)

9. Primary Outcome: Tmax Whole Blood Total Radioactivity of Radiolabelled Prucalopride Succinate
Time Frame: Over 240 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Median (Full Range); unit: hours
Arm/Group | [14C] PRUCALOPRIDE SUCCINATE
Number analyzed (Participants) | 6
hours | 2.75 [1.53 to 4.00]

10. Primary Outcome: Half-Life Whole Blood Total Radioactivity of Radiolabelled Prucalopride Succinate
Time Frame: Over 240 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | [14C] PRUCALOPRIDE SUCCINATE
Number analyzed (Participants) | 6
hours | 18.0 (5.18)

11. Primary Outcome: AUC 0→∞ Plasma Total Radioactivity of Radiolabelled Prucalopride Succinate
Time Frame: Over 240 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: ng equivalents*h/ml
Arm/Group | [14C] PRUCALOPRIDE SUCCINATE
Number analyzed (Participants) | 6
ng equivalents*h/ml | 102 (11.2)

12. Primary Outcome: Cmax Plasma Total Radioactivity of Radiolabelled Prucalopride Succinate
Time Frame: Over 240 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: ng equivalents/ml
Arm/Group | [14C] PRUCALOPRIDE SUCCINATE
Number analyzed (Participants) | 6
ng equivalents/ml | 4.14 (1.29)

13. Primary Outcome: Tmax Plasma Total Radioactivity of Radiolabelled Prucalopride Succinate
Time Frame: Over 240 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Median (Full Range); unit: hours
Arm/Group | [14C] PRUCALOPRIDE SUCCINATE
Number analyzed (Participants) | 6
hours | 2.25 [1.13 to 4.00]

14. Primary Outcome: Half-Life Plasma Total Radioactivity of Radiolabelled Prucalopride Succinate
Time Frame: Over 240 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | [14C] PRUCALOPRIDE SUCCINATE
Number analyzed (Participants) | 6
hours | 19.7 (5.64)

15. Primary Outcome: Percent Total Radioactivity Excreted in Urine of Radiolabelled Prucalopride Succinate
Time Frame: 240 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: percentage of radioactvity
Arm/Group | [14C] PRUCALOPRIDE SUCCINATE
Number analyzed (Participants) | 6
percentage of radioactvity | 84.2 (8.88)

16. Primary Outcome: Percent Total Radioactivity Excreted in Stool of Radiolabelled Prucalopride Succinate
Time Frame: Over 240 hours post-dose
Population: Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: percentage of radioactivity
Arm/Group | [14C] PRUCALOPRIDE SUCCINATE
Number analyzed (Participants) | 6
percentage of radioactivity | 13.3 (1.73)

ADVERSE EVENTS:
Arm/Group | [14C] PRUCALOPRIDE SUCCINATE
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | [14C] PRUCALOPRIDE SUCCINATE (N=6)
Abdominal discomfort (Gastrointestinal disorders) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (6)
Presyncope (Nervous system disorders) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.